CLINICAL TRIAL: NCT03540290
Title: Treatment of Peri-implant Mucositis by Means of Implant Decontamination and Modification of the Implant Supported-prosthesis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Beatriz de Tapia, Clinical professor, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2017-01
Record Dates: First submitted 2018-04-27; First posted 2018-05-30 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical instrumentation and oral hygiene instructions (Active Comparator)
  Interventions: Procedure: Modification of the implant supported prostheses in order to facilitate oral hygiene
- Modification of the implant supported prostheses (Experimental)
  Interventions: Procedure: Modification of the implant supported prostheses in order to facilitate oral hygiene

INTERVENTIONS:
Procedure: Modification of the implant supported prostheses in order to facilitate oral hygiene — Peri-implant mucositis will be treated by individualized oral hygiene instructions and decontamination of the implant surface by ultrasonic device with a plastic tip and plastic curettes plus the modification of the implant prosthesis in order to facilitate oral hygiene access

SUMMARY:
To test the modification of the implant prosthesis, in order to facilitate access to biofilm control, in combination with decontamination of the implant surface by means of an ultrasonic device with a plastic tip and plastic curettes, in comparison with the decontamination of the implant surface by means of an ultrasonic device with a plastic tip and plastic curettes, and no modification of the implant prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* (1) Presence of, at least, one titanium implant exhibiting peri-implant mucositis, defined as bleeding on gentle probing (0.15 N) in at least one peri-implant site.

  (2) No signs of loss of supporting bone after initial bone remodelling. In cases where baseline radiograph is available, it will be used for comparison, otherwise a maximum of 2 mm of crestal bone loss will be accepted (5).

  (3) Single tooth and bridgework restoration with an inappropriate prosthesis design or contour which difficult oral hygiene access (overcontoured prosthesis, prostheses presenting closed embrasures, an abrupt emergence profile or excessive buccal flanges).

  (4) Presence of >1 mm of keratinized peri-implant mucosa.

  (5) A good level of oral hygiene, defined as an O'Leary et al. plaque index <25% (16).

  (6) Absence of systemic diseases that could influence the outcome of the therapy (i.e. controlled diabetes, with HbA1c<7, patients will be included).

  (7) Non-smoker or light smoking status in smokers (<10 cigarettes/day).

Exclusion Criteria:

* (1) Untreated periodontal conditions.

  (2) Pregnant or lactating women.

  (3) Patients who received systemic antibiotics in the last 3 months.

  (4) Patients who received treatment of PM in the past 3 months.

  (5) Patients receiving corticoids or medications known to have effect on gingival growth i.e. calcium channel antagonists, immunosuppressants or antiepileptic drugs.

In those cases diagnosed with peri-implantitis, individualized treatment will be provided, apart from the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-01-10 (Actual); Primary Completion 2018-12-12 (Estimated); Study Completion 2019-06-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate modified sulcus Bleeding Index changes at 3 and 6 months, by the modification of the implant prosthesis in order to facilitate oral hygiene, hygiene instructions and surface decontamination | 1, 3 and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Sant Cugat Del Vallès, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The results obtained are expected to be published in both national and international journals. In addition, the results will be disseminated national and international scientific events.